CLINICAL TRIAL: NCT03972488
Title: A Phase III Multi-center, Randomized, Open-label Study to Evaluate the Efficacy and Safety of Lutathera in Patients With Grade 2 and Grade 3 Advanced GEP-NET
Brief Title: Study to Evaluate the Efficacy and Safety of Lutathera in Patients With Grade 2 and Grade 3 Advanced GEP-NET
Acronym: NETTER-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CAAA601A22301; 2023-507443-10-00 (Other: EU CTIS)
Record Dates: First submitted 2019-05-24; First posted 2019-06-03 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Gastro-enteropancreatic Neuroendocrine Tumor
Keywords: Lutathera; GEP-NET; NETTER-2; 177Lu-DOTA0-TATE; Lutetium oxodotreotide; Lutetium dotatate; AAA601
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor | interventions — lutetium Lu 177 dotatate; Receptor-Like Protein Tyrosine Phosphatases, Class 2; Octreotide; pasireotide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Lutathera® plus Octreotide LAR 30 mg (Investigational arm) (Experimental): Lutathera treatment consisted of a cumulative administered radioactivity of 29.6 GBq (800mCi) (7.4 GBq/200 mCi x 4 administrations every 8 +/- 1 week). Participants in the Lutathera arm were concomitantly administered with octreotide LAR 30 mg (Sandostatin LAR Depot) the day after each administration of Lutathera and no earlier than 4 hours after completion of the Lutathera infusion. Once Lutathera treatment completed, participants continued the 4-week interval administrations of 30 mg octreotide LAR until the completion of the Treatment Phase. Concomitantly with Lutathera, sterile amino acid solution was administered to minimize renal radiation exposure during Lutathera treatment.
  Interventions: Drug: Lutathera; Drug: 30 mg Octreotide long acting repeatable (LAR) (Sandostatin LAR Depot); Drug: 2.5% Lys-Arg sterile amino acid solution
- Octreotide LAR 60 mg (Control arm) (Active Comparator): Participants were administered with octreotide LAR 60 mg (Sandostatin LAR Depot) at 4-week intervals until the completion of the Treatment Phase.
  Interventions: Drug: High dose 60 mg octreotide long-acting repeatable
- Optional post-progression re-treatment with Lutathera (Experimental): Participants who received Lutathera in experimental arm and who progressed and met re-treatment eligibility criteria received additional 2 - 4 cycles of Lutathera (7.4 GBq/200 mCi x 4 cycles)
  Interventions: Drug: Lutathera
- Optional post-progression cross-over to Lutathera (Active Comparator): Participants who received Octreotide LAR in Active comparator arm and who progressed and met cross-over eligibility criteria received maximum 4 cycles of Lutaathera (7.4 GBq/200 mCi x 4 cycles) plus octreotide long-acting (30 mg every 8 weeks).
  Interventions: Drug: Lutathera
- Optional post-progression re-treatment with Lutathera after cross-over (Active Comparator): Participants who received Octreotide LAR in Active comparator arm subsequently entered cross-over, received Lutathera in cross-over, progressed for the second time and met re-treatment eligibility criteria could receive additional 2 - 4 cycles of Lutathera (7.4 GBq/200 mCi x 4 cycles).
  Interventions: Drug: Lutathera; Drug: High dose 60 mg octreotide long-acting repeatable

INTERVENTIONS:
Drug: Lutathera — Lutathera is a sterile radiopharmaceutical supplied as a ready-to-use solution for infusion containing 177Lu-DOTA0-Tyr3-octreotate as a drug substance with a volumetric activity of 370 MBq/mL at reference date and time (calibration time). Each Lutathera infusion continued for 30 min.
  Other Names: AAA601
  Arms: Lutathera® plus Octreotide LAR 30 mg (Investigational arm); Optional post-progression cross-over to Lutathera; Optional post-progression re-treatment with Lutathera; Optional post-progression re-treatment with Lutathera after cross-over
Drug: 30 mg Octreotide long acting repeatable (LAR) (Sandostatin LAR Depot) — Sandostatin® LAR Depot (octreotide LAR) is a pharmaceutical that was available in single-use kits containing a 6-mL vial of 10 mg, 20 mg, or 30 mg strength for intramuscular injection, a syringe containing 2.5 mL of diluent, two sterile 1½" 19-gauge needles, and two alcohol wipes.
  Other Names: SOM230
  Arms: Lutathera® plus Octreotide LAR 30 mg (Investigational arm)
Drug: 2.5% Lys-Arg sterile amino acid solution — Participants who received Lutathera were administered a concomitant 2.5% Lys-Arg solution for kidney protection, with each Lutathera dose. The 2.5% Lys-Arg solution was administered intravenously for 4 hours (infusion rate: 250 ml/h); the infusion was to start 30 minutes prior to the start of the Lutathera infusion and continue during (30 min) and up to at least 3 hours after the Lutathera infusion.
  Arms: Lutathera® plus Octreotide LAR 30 mg (Investigational arm)
Drug: High dose 60 mg octreotide long-acting repeatable — Sandostatin® LAR Depot (octreotide LAR) is a pharmaceutical that was available in single-use kits containing a 6-mL vial of 10 mg, 20 mg, or 30 mg strength for intramuscular injection, a syringe containing 2.5 mL of diluent, two sterile 1½" 19-gauge needles, and two alcohol wipes.
  Arms: Octreotide LAR 60 mg (Control arm); Optional post-progression re-treatment with Lutathera after cross-over

SUMMARY:
The aim of NETTER-2 was to determine if Lutathera in combination with long-acting octreotide prolongs progression free survival (PFS) in gastroenteropancreatic neuroendocrine tumor (GEP-NET) patients with high proliferation rate tumors (G2 and G3), when given as a first line treatment compared to treatment with high dose (60 mg) long-acting octreotide. Somatostatin analog (SSA) naive patients were eligible, as well as patients previously treated with SSAs in the absence of progression.

DETAILED DESCRIPTION:
The study consisted of a screening phase, a treatment phase, an optional cross-over phase for subjects assigned to the control arm, optional re-treatment phase for subjects assigned to the Lutathera arm, and a follow-up phase. This study compared treatment with Lutathera (7.4 GBq/200 mCi 4 × administrations every 8 weeks ± 1 week; cumulative dose: 29.6 GBq/800mCi) plus octreotide long-acting release (LAR) (30 mg every 8 weeks during Lutathera treatment and every 4 weeks after last Lutathera treatment) and high dose octreotide LAR (60 mg every 4 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Presence of metastasized or locally advanced, inoperable (curative intent) histologically proven, well differentiated Grade 2 or Grade 3 gastroenteropancreatic neuroendocrine (GEP-NET) tumor diagnosed within 6 months prior to screening.
* Ki67 index ≥10 and ≤ 55%
* Patients ≥ 15 years of age and a body weight of > 40 kg at screening
* Expression of somatostatin receptors on all target lesions documented by CT/MRI scans, assessed by any of the following somatostatin receptor imaging (SRI) modalities within 3 months prior to randomization: [68Ga]-DOTA-TOC (e.g. Somakit-TOC®) PET/CT (or MRI when applicable based on target lesions) imaging, [68Ga]-DOTA-TATE PET/CT (or MRI when applicable based on target lesions) imaging (e.g. NETSPOT®), Somatostatin Receptor scintigraphy (SRS) with [111In]-pentetreotide (Octreoscan® SPECT/CT), SRS with [99mTc]-Tektrotyd, [64Cu]-DOTA-TATE PET/CT (or MRI when applicable based on target lesions) imaging.
* The tumor uptake observed in the target lesions must be > normal liver uptake.
* Karnofsky Performance Score (KPS) ≥ 60
* Presence of at least 1 measurable site of disease
* Patients who have provided a signed informed consent form to participate in the study, obtained prior to the start of any protocol related activities

Exclusion Criteria:

* Creatinine clearance < 40 mL/min calculated by the Cockroft Gault method
* Hb concentration < 5.0 mmol/L (<8.0 g/dL); WBC < 2x10E9/L (2000/mm3); platelets < 75x10E9/L (75x10E3/mm3)
* Total bilirubin > 3 x ULN
* Serum albumin < 3.0 g/dL unless prothrombin time is within the normal range
* Pregnancy or lactation
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, are not allowed to participate in this study UNLESS they are using highly effective methods of contraception throughout the study treatment period (including cross-over and re-treatment, if applicable) and for 7 months after study drug discontinuation
* Peptide receptor radionuclide therapy (PRRT) at any time prior to randomization in the study.
* Documented RECIST progression to previous treatments for the current GEP-NET at any time prior to randomization
* Patients for whom in the opinion of the investigator other therapeutic options (eg chemo-, targeted therapy) are considered more appropriate than therapy offered in the study, based on patient and disease characteristics
* Any previous therapy with Interferons, Everolimus (mTOR-inhibitors), chemotherapy or other systemic therapies for GEP-NET administered for more than 1 month or within 12 weeks prior to randomization in the study.
* Any previous radioembolization, chemoembolization and radiofrequency ablation for GEP-NET
* Any surgery within 12 weeks prior to randomization in the study
* Known brain metastases, unless these metastases have been treated and stabilized for at least 24 weeks, prior to screening in the study. Patients with a history of brain metastases must have a head CT or MRI with contrast to document stable disease prior to randomization in the study.
* Uncontrolled congestive heart failure (NYHA II, III, IV). Patients with history of congestive heart failure who do not violate this exclusion criterion will undergo an evaluation of their cardiac ejection fraction prior to randomization via echocardiography. The results from an earlier assessment (not exceeding 30 days prior to randomization) may substitute the evaluation at the discretion of the Investigator, if no clinical worsening is noted. The patient's measured cardiac ejection fraction in these patients must be ≥40% before randomization.
* QTcF > 470 msec for females and QTcF > 450 msec for males or congenital long QT syndrome
* Uncontrolled diabetes mellitus as defined by hemoglobin A1c value > 7.5%
* Hyperkaleamia > 6.0 mmol/L (CTCAE Grade 3) which is not corrected prior to study enrolment
* Any patient receiving treatment with short-acting octreotide, which cannot be interrupted for 24 h before and 24 h after the administration of Lutathera, or any patient receiving treatment with SSAs (e.g. octreotide long-acting), which cannot be interrupted for at least 6 weeks before the administration of Lutathera.
* Patients with any other significant medical, psychiatric, or surgical condition, currently uncontrolled by treatment, which may interfere with the completion of the study.
* Prior external beam radiation therapy to more than 25% of the bone marrow.
* Current spontaneous urinary incontinence
* Other known co-existing malignancies except non-melanoma skin cancer and carcinoma in situ of the uterine cervix, unless definitively treated and proven no evidence of recurrence for 5 years
* Patient with known incompatibility to CT Scans with IV contrast due to allergic reaction or renal insufficiency. If such a patient can be imaged with MRI, then the patient would not be excluded.
* Hypersensitivity to any somatostatin analogues, the IMPs active substance or to any of the excipients.
* Patients who have participated in any therapeutic clinical study/received any investigational agent within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2027-10-29 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (40):
- United States (6):
  - Yale Cancer Center, New Haven, Connecticut
  - USF - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Iowa Hospitals and Clinics - Oncology, Iowa City, Iowa
  - University of Kentucky UK Markey Cancer Center, Lexington, Kentucky
  - Mayo Clinic - Oncology, Rochester, Minnesota
  - MD Anderson Cancer Center, Houston, Texas
- Canada (4):
  - London Health Sciences Centre, University of Western Ontario - Oncology, London
  - Centre Hospitalier Universitaire de Quebec, Québec
  - Sunnybrook Health Sciences Centre, Toronto
  - BC Cancer Agency, Vancouver
- France (5):
  - CHU Paris Nord-Val de Seine, Clichy
  - Hospices Civils de Lyon (HCL) - Hopital Edouard Herriot, Lyon
  - Institut du Cancer de Montpellier - Oncology, Montpellier
  - CHU-Hôtel Dieu Service de Médecine Nucléaire, Nantes
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen - Klinik für Nuklearmedizin, Essen
- Italy (8):
  - A.O.di Bologna Policl.S.Orsola, Bologna
  - University of Genova - Oncology, Genova
  - Istituto Oncologico Romagnolo, Meldola
  - Fondazione Irccs Istituto Nazionale Tumori, Milan
  - Ieo, Irccs, Milan
  - IRCCS fondazione Pascale - Oncology, Napoli
  - Arcispedale Santa Maria Nuova, Reggio Emilia - Oncology, Reggio Emilia
  - Azienda Ospedaliera Sant'Andrea - Università La Sapienza U.O.C. Mal App. Digerente e - Oncology, Roma
- Netherlands (2):
  - Erasmus Medisch Centrum, Rotterdam
  - UMC Utrecht - Oncology, Utrecht
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center - Oncology, Seoul
  - Seoul National University Hospital - Department of Internal Medicine, Seoul
  - Severance Hospital, Yonsei University Health System - Medical Oncology, Seoul
- Spain (4):
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (5):
  - Bristol Haematology and Oncology Centre, Bristol
  - Guys And St Thomas Hospital, London
  - Kings College Hospital - Oncology, London
  - Royal Free Hospital, London, London
  - Weston Park Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Result] Singh S, Halperin D, Myrehaug S, Herrmann K, Pavel M, Kunz PL, Chasen B, Tafuto S, Lastoria S, Capdevila J, Garcia-Burillo A, Oh DY, Yoo C, Halfdanarson TR, Falk S, Folitar I, Zhang Y, Aimone P, de Herder WW, Ferone D; all the NETTER-2 Trial Investigators. [177Lu]Lu-DOTA-TATE plus long-acting octreotide versus high-dose long-acting octreotide for the treatment of newly diagnosed, advanced grade 2-3, well-differentiated, gastroenteropancreatic neuroendocrine tumours (NETTER-2): an open-label, randomised, phase 3 study. Lancet. 2024 Jun 29;403(10446):2807-2817. doi: 10.1016/S0140-6736(24)00701-3. Epub 2024 Jun 5. PMID 38851203
- [Derived] Bahri N, Crook C, Daneng Li. Casting a Wide NET: When Is the Optimal Time for 177Lu-Dotatate Treatment? Oncology (Williston Park). 2024 Nov 5;38(11):442-443. doi: 10.46883/2024.25921029. PMID 39570708
- [Derived] Jungels C, Deleporte A. State of the art and future directions in the systemic treatment of neuroendocrine neoplasms. Curr Opin Oncol. 2021 Jul 1;33(4):378-385. doi: 10.1097/CCO.0000000000000740. PMID 33973550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study randomized subjects in 38 centers in 9 participating countries. Overall, 222 subjects were planned to be randomized (2:1) to Lutathera arm or control arm.
Period: Overall Study
Arm/Group | Lutathera® Plus Octreotide LAR 30 mg (Investigational Arm) | Octreotide LAR 60 mg (Control Arm)
Started | 151 | 75
Participants Treated in Treatment Period | 147 | 73
Participants Not Treated in Treatment Period | 4 | 2
Participants Entered Crossover Treatment Period | 0 | 29
Participants Entered Retreatment Period | 8 | 0
Completed (Completed = Treatment ongoing) | 78 | 15
Not Completed | 73 | 60
Not completed — Progressive disease | 42 | 44
Not completed — Physician Decision | 13 | 7
Not completed — Adverse Event | 8 | 1
Not completed — Death | 4 | 4
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Other = untreated or stopped treatment by patient decision but agreed to be followed-up | 3 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) comprises all participants to whom study treatment has been assigned by randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lutathera® Plus Octreotide LAR 30 mg (Investigational Arm) | Octreotide LAR 60 mg (Control Arm) | Total
Number analyzed (Participants) | 151 | 75 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (13.21) | 59.6 (11.52) | 60.0 (12.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 35 | 105
  Male | 81 | 40 | 121
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 115 | 50 | 165
  Black or African American | 3 | 2 | 5
  Asian (Indian & Korean) | 23 | 11 | 34
  American Indian or Alaska Native | 1 | 0 | 1
  Multiple | 1 | 0 | 1
  Missing | 8 | 12 | 20

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Per Central Assessment
Description: PFS is the time from randomization to the first line progression (centrally assessed according to RECIST 1.1) or death due to any cause. Progression is defined using Response Evaluation Criteria in Solid Tumor Criteria (RECIST 1.1) as a 20% increase in the sum of diameters of all measured target lesions or unequivocal progression of non-target lesions or appearance of a new lesion.
Time Frame: from randomization to the first line progression or death due to any cause, up to approx. 42 months
Population: Full Analysis Set (FAS) comprises all participants to whom study treatment has been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lutathera® Plus Octreotide LAR 30 mg (Investigational Arm) | Octreotide LAR 60 mg (Control Arm)
Number analyzed (Participants) | 151 | 75
months | 22.8 [19.4 to NA] — NA: The upper limit of CI was not reached because of insufficient number of participants with events in the Lutathera arm | 8.5 [7.7 to 13.8]
Statistical Analysis 1: Comparison: Lutathera® Plus Octreotide LAR 30 mg (Investigational Arm) vs Octreotide LAR 60 mg (Control Arm); Test type: Superiority; p < 0.0001, Log Rank; Stratified one-sided P-value; Hazard Ratio (HR) = 0.276, 95% CI 2-sided [0.182 to 0.418]

2. Secondary Outcome: Overall Response Rate (ORR) Per Central Assessment (Key Secondary)
Description: ORR is defined as the percentage of patients with the best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1. CR = Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR = At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approx. 42 months
Population: FAS comprises all participants to whom study treatment has been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lutathera® Plus Octreotide LAR 30 mg (Investigational Arm) | Octreotide LAR 60 mg (Control Arm)
Number analyzed (Participants) | 151 | 75
Percentage of participants | 43.0 [35.0 to 51.3] | 9.3 [3.8 to 18.3]
Statistical Analysis 1: Comparison: Lutathera® Plus Octreotide LAR 30 mg (Investigational Arm) vs Octreotide LAR 60 mg (Control Arm); Test type: Superiority; p < 0.0001, Stratified One-sided p-value; Stratified Odds Ratio = 7.81, 95% CI 2-sided [3.32 to 18.40]

3. Secondary Outcome: Time to Deteriration (TTD) Global Health Status, Diarrhea, Fatigue, Pain (EORTC QLQ-C30) (Key Secondary)
Description: TTD is defined as the first deterioration of at least 10 points from baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30): global health status, diarrhea, fatigue, and pain.
  The Quality of Life Questionnaire C30 (QLQ-C30) was developed by the European Organization for Research and Treatment of Cancer (EORTC) to assess quality of life in cancer patients. It includes five function domains (physical, emotional, social, role, cognitive), eight symptoms (fatigue, pain, nausea/vomiting, constipation, diarrhea, insomnia, dyspnea, and appetite loss), as well as global health/quality-of-life and financial impact. Subjects respond on a four-point scale from "not at all" to "very much" for most items. Raw scores are linearly transformed so each score ranged a 0-100, where higher scores indicate worse symptoms (e.g., more severe/worsened) and lower scores indicate less symptoms (e.g., less severe/improvement).
Time Frame: Up to approx. 42 months
Population: FAS comprises all participants to whom study treatment has been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lutathera® Plus Octreotide LAR 30 mg (Investigational Arm) | Octreotide LAR 60 mg (Control Arm)
Number analyzed (Participants) | 151 | 75
months
  Global Health status | 13.2 [8.8 to 17.2] | 8.6 [5.8 to 14.0]
  Diarrhea | 17.4 [14.4 to 28.2] | 17.3 [8.1 to NA] — NA: The upper limit of CI was not reached because of insufficient number of participants with events in the Octreotide arm
  Fatigue | 6.0 [3.4 to 6.8] | 6.0 [3.9 to 11.0]
  Pain | 10.3 [6.0 to 13.6] | 8.6 [3.9 to 13.7]
Statistical Analysis 1: Comparison: Lutathera® Plus Octreotide LAR 30 mg (Investigational Arm) vs Octreotide LAR 60 mg (Control Arm); Global Health Status; Test type: Superiority; p = 0.2222, Log Rank; Stratified one-sided P-value; Hazard Ratio (HR) = 0.856, 95% CI 2-sided [0.570 to 1.283]

4. Secondary Outcome: Disease Control Rate (DCR) Per Central Assessment
Description: Disease Control Rate is the percentage of participants with a best overall response of complete response (CR), partial response (PR) or stable disease (SD) (centrally assessed according to RECIST 1.1). CR = Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR = At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters; SD = Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease (PD).
Time Frame: Up to approx. 42 months
Population: FAS comprises all participants to whom study treatment has been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lutathera® Plus Octreotide LAR 30 mg (Investigational Arm) | Octreotide LAR 60 mg (Control Arm)
Number analyzed (Participants) | 151 | 75
Percentage of participants | 90.7 [84.9 to 94.8] | 66.7 [54.8 to 77.1]

5. Secondary Outcome: Duration of Response (DOR) Per Central Assessment
Description: Duration of Response defined as time from first complete or partial response to progression or death due to underlying cancer according to RECIST 1.1.
Time Frame: Up to approx. 42 months
Population: FAS comprises all participants to whom study treatment has been assigned by randomization. Only participants who had a response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lutathera® Plus Octreotide LAR 30 mg (Investigational Arm) | Octreotide LAR 60 mg (Control Arm)
Number analyzed (Participants) | 65 | 7
months | 23.3 [18.4 to NA] — NA: The upper limit of CI was not reached because of insufficient number of participants with events in the Lutathera arm | NA [NA to NA] — NA: The median was not reached because of insufficient number of participants with events in the Octreotide arm

6. Secondary Outcome: Rate of Adverse Events
Description: Rate of adverse events scored according to CTCAE grade
Time Frame: from FPFV until end of study (about 94 months)
Reporting Status: Not Posted, anticipated posting 2028-10

7. Secondary Outcome: Rate of Laboratory Toxicities
Description: Rate of laboratory toxicities scored according to CTCAE grade
Time Frame: from FPFV until end of study (about 94 months)
Reporting Status: Not Posted, anticipated posting 2028-10

8. Secondary Outcome: Overall Survival (OS)
Description: OS is the time from randomization date until day of death due to any cause.
Time Frame: from FPFV until end of study (about 94 months)
Reporting Status: Not Posted, anticipated posting 2028-10

ADVERSE EVENTS:
Time Frame: On-treatment AEs and deaths were collected from the first dose of study treatment up to 30 days after last dose of study medication, up to 42 months.
Description: Any sign or symptom that occurs during the conduct of the trial.
Groups:
- Lutathera® Plus Octreotide LAR 30 mg: Lutathera treatment consisted of a cumulative administered radioactivity of 29.6 GBq (800mCi) (7.4 GBq/200 mCi x 4 administrations every 8 +/- 1 week). Participants in the Lutathera arm were concomitantly administered with octreotide LAR 30 mg (Sandostatin LAR Depot) the day after each administration of Lutathera and no earlier than 4 hours after completion of the Lutathera infusion. Once Lutathera treatment completed, participants continued the 4-week interval administrations of 30 mg octreotide LAR until the completion of the Treatment Phase. Concomitantly with Lutathera, sterile amino acid solution was administered to minimize renal radiation exposure during Lutathera treatment.
- Crossover Lutathera: Participants who received Octreotide LAR in Active comparator Arm and who progressed and met cross over eligibility criteria received maximum 4 cycles of Lutathera (7.4 GBq/200 mCi x 4 cycles) plus octreotide long-acting (30 mg every 8 weeks)
- Re-Treatment Lutathera: Participants who received Lutathera in experimental arm and who progressed and met re treatment eligibility criteria received additional 2-4 cycles of Lutathera (7.4 GBq/200 mCi x 4 cycles)
Arm/Group | Lutathera® Plus Octreotide LAR 30 mg | Octreotide LAR 60 mg (Control Arm) | Crossover Lutathera | Re-Treatment Lutathera
All-Cause Mortality (participants affected / at risk) | 32/147 | 14/73 | 3/29 | 0/8
Serious Adverse Events (participants affected / at risk) | 30/147 | 15/73 | 2/29 | 0/8
Other Adverse Events (participants affected / at risk) | 129/147 | 65/73 | 22/29 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lutathera® Plus Octreotide LAR 30 mg (N=147) | Octreotide LAR 60 mg (Control Arm) (N=73) | Crossover Lutathera (N=29) | Re-Treatment Lutathera (N=8)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Carcinoid heart disease (Cardiac disorders) | 0 | 1 | 0 | 0
Pulmonary valve disease (Cardiac disorders) | 1 | 0 | 0 | 0
Carcinoid syndrome (Endocrine disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 5 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 1 | 0 | 0
Infusion site extravasation (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Gallbladder rupture (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0
Waist circumference increased (Investigations) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lutathera® Plus Octreotide LAR 30 mg (N=147) | Octreotide LAR 60 mg (Control Arm) (N=73) | Crossover Lutathera (N=29) | Re-Treatment Lutathera (N=8)
Anaemia (Blood and lymphatic system disorders) | 27 | 4 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 9 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 12 | 6 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 24 | 20 | 6 | 0
Abdominal pain upper (Gastrointestinal disorders) | 11 | 6 | 3 | 0
Constipation (Gastrointestinal disorders) | 15 | 6 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 38 | 25 | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 7 | 1 | 1 | 1
Flatulence (Gastrointestinal disorders) | 11 | 4 | 1 | 0
Nausea (Gastrointestinal disorders) | 39 | 13 | 8 | 3
Vomiting (Gastrointestinal disorders) | 21 | 6 | 2 | 1
Asthenia (General disorders) | 28 | 9 | 0 | 2
Fatigue (General disorders) | 29 | 13 | 7 | 0
Injection site pain (General disorders) | 4 | 4 | 0 | 0
Oedema peripheral (General disorders) | 17 | 5 | 1 | 0
Pain (General disorders) | 1 | 0 | 1 | 1
Pyrexia (General disorders) | 11 | 3 | 0 | 0
COVID-19 (Infections and infestations) | 28 | 10 | 1 | 0
Alanine aminotransferase increased (Investigations) | 16 | 10 | 4 | 0
Aspartate aminotransferase increased (Investigations) | 16 | 8 | 4 | 0
Blood alkaline phosphatase increased (Investigations) | 7 | 4 | 2 | 0
Blood bilirubin increased (Investigations) | 4 | 5 | 0 | 0
Blood creatinine increased (Investigations) | 9 | 2 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 12 | 4 | 1 | 0
Creatinine renal clearance decreased (Investigations) | 1 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 12 | 8 | 2 | 0
Lymphocyte count decreased (Investigations) | 16 | 0 | 2 | 0
Neutrophil count decreased (Investigations) | 9 | 0 | 0 | 0
Platelet count decreased (Investigations) | 24 | 4 | 1 | 1
Weight decreased (Investigations) | 14 | 2 | 0 | 1
Weight increased (Investigations) | 18 | 5 | 3 | 0
White blood cell count decreased (Investigations) | 19 | 3 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 19 | 7 | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 20 | 10 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 6 | 1 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 4 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 6 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 7 | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 4 | 0 | 0
Dizziness (Nervous system disorders) | 12 | 3 | 4 | 0
Headache (Nervous system disorders) | 16 | 5 | 3 | 1
Insomnia (Psychiatric disorders) | 11 | 3 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 1 | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 4 | 1 | 0
Menopause (Social circumstances) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 7 | 4 | 1 | 0
Hypertension (Vascular disorders) | 13 | 5 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e., data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT03972488/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT03972488/SAP_001.pdf